CLINICAL TRIAL: NCT04956588
Title: A Multicenter, Randomized, Single-blind, Parallel-controlled Clinical Trial to Evaluate the Safety and Efficacy of Smart Orthopedic Minimally Invasive Surgical Systems for Spinal Surgery
Brief Title: Evaluation of the Safety and Efficacy of Smart Orthopedic Minimally Invasive Surgical Systems for Spinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2017079
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Spine Disease; Spinal Fractures
Keywords: smart orthopedics; minimally invasive surgical systems; spinal surgery
MeSH Terms: conditions — Spinal Diseases; Spinal Fractures | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded when evaluating the subject's imaging data (i.e., when calculating the deviation of the nail placement).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Combination Product: surgical robot
- control group (Active Comparator)
  Interventions: Combination Product: controlled approach

INTERVENTIONS:
Combination Product: surgical robot — The surgical robot completed the screw placement according to the surgical plan, and the researchers closely monitored the screw placement process.
  Arms: experimental group
Combination Product: controlled approach — The screw placement was performed using a controlled approach according to the surgical plan.
  Arms: control group

SUMMARY:
To evaluate the safety and effectiveness of the intelligent orthopedic minimally invasive surgery system developed by Shenzhen Xinjunte Intelligent Medical Equipment Co., Ltd. in spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-65, gender unlimited; In line with the surgical conditions for spinal surgery requiring Kirschner wire implantation, and the treatment plan allows open or minimally invasive surgery; Signed the informed consent and agreed to participate in the study; Complete the filter check and meet all the entry criteria in the filter table.

Exclusion Criteria:

- Subject meeting the exclusion criteria; People with metal allergy; Women who are lactating or pregnant, and the possibility of pregnancy cannot be ruled out; Subjects with coagulation dysfunction; Subjects who have failed spinal surgery and need a second operation; Subjects with spinal tumors, deformities and slippery vertebrae; Candidates who have participated in clinical trials related to other drugs and medical devices within the past 3 months; Any other circumstances in which the Investigator deems it inappropriate to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incorrect placement of guide pin | During operation
  After the subject completes the preparation for guide needle placement (e.g. reduction), a C-arm scan is performed. Get the image. Surgical planning is performed on images. Control robot positioning. The doctor completes the insertion of the guide needle. Then the C-arm scan image was obtained again. Fusion of two groups of images on a third-party software. The deviation distance between the entry and exit points of the guide needle and the surgical plan was measured. The accuracy of guide needle placement was evaluated by the deviation of guide needle placement.
Number of X-ray exposures | During operation
  The number of exposures was defined as the number of times the investigator used the X-ray during the operative period and also included the number of exposures performed to determine the surgical site.
X-ray exposure time | During operation
  X-ray exposure time refers to the total time of using X-rays from the planning of the operation to the end of the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No